CLINICAL TRIAL: NCT06642558
Title: A Phase I/II, Single Center, Randomized, Double-Blinded, Placebo-Controlled Clinical Trial to Evaluate the Safety and Immunogenicity of Recombinant Respiratory Syncytial Virus Vaccine (CHO Cell) in Healthy Subjects Aged 18 Years and Above
Brief Title: Safety and Immunogenicity of Recombinant RSV Vaccine (CHO Cell) in Healthy Subjects Aged 18 Years and Above
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: MAXVAX Biotechnology Limited Liability Company (Industry)
Collaborators: Henan Center for Disease Control and Prevention (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MKKCT-900-001
Record Dates: First submitted 2024-10-11; First posted 2024-10-15 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Respiratory Syncytial Virus (RSV)
MeSH Terms: interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (12):
- Low dose vaccine group in subjects aged 18-59 years - Phase 1 (Experimental): Subjects aged 18-59 years in phase 1 will receive single dose of Recombinant Respiratory Syncytial Virus Vaccine (CHO Cells)(low dose), by IM injection into the deltoid region of the arm.
  Interventions: Biological: Recombinant Respiratory Syncytial Virus Vaccine (CHO Cells)(low dose)
- High dose vaccine group in subjects aged 18-59 years - Phase 1 (Experimental): Subjects aged 18-59 years in phase 1 will receive single dose of Recombinant Respiratory Syncytial Virus Vaccine (CHO Cells)(high dose), by IM injection into the deltoid region of the arm.
  Interventions: Biological: Recombinant Respiratory Syncytial Virus Vaccine (CHO Cells)(high dose)
- Placebo group in subjects aged 18-59 years - Phase 1 (Placebo Comparator): Subjects aged 18-59 years in phase 1 will receive single dose of placebo, by IM injection into the deltoid region of the arm.
  Interventions: Biological: Placebo (Saline solution)
- Low dose vaccine group in subjects aged ≥60 years - Phase 1 (Experimental): Subjects aged ≥60 years in phase 1 will receive single dose of Recombinant Respiratory Syncytial Virus Vaccine (CHO Cells)(low dose), by IM injection into the deltoid region of the arm.
  Interventions: Biological: Recombinant Respiratory Syncytial Virus Vaccine (CHO Cells)(low dose)
- High dose vaccine group in subjects aged ≥60 years - Phase 1 (Experimental): Subjects aged ≥60 years in phase 1 will receive single dose of Recombinant Respiratory Syncytial Virus Vaccine (CHO Cells)(high dose), by IM injection into the deltoid region of the arm.
  Interventions: Biological: Recombinant Respiratory Syncytial Virus Vaccine (CHO Cells)(high dose)
- Placebo group in subjects aged ≥60 years - Phase 1 (Placebo Comparator): Subjects aged ≥60 years in phase 1 will receive single dose of placebo, by IM injection into the deltoid region of the arm.
  Interventions: Biological: Placebo (Saline solution)
- Low dose vaccine group in subjects aged 50-59 years - Phase 2 (Experimental): Subjects aged 50-59 years in phase 2 will receive single dose of Recombinant Respiratory Syncytial Virus Vaccine (CHO Cells)(low dose), by IM injection into the deltoid region of the arm.
  Interventions: Biological: Recombinant Respiratory Syncytial Virus Vaccine (CHO Cells)(low dose)
- High dose vaccine group in subjects aged 50-59 years - Phase 2 (Experimental): Subjects aged 50-59 years in phase 2 will receive single dose of Recombinant Respiratory Syncytial Virus Vaccine (CHO Cells)(high dose), by IM injection into the deltoid region of the arm.
  Interventions: Biological: Recombinant Respiratory Syncytial Virus Vaccine (CHO Cells)(high dose)
- Placebo group in subjects aged 50-59 years - Phase 2 (Placebo Comparator): Subjects aged 50-59 years in phase 2 will receive single dose of placebo, by IM injection into the deltoid region of the arm.
  Interventions: Biological: Placebo (Saline solution)
- Low dose vaccine group in subjects aged ≥60 years - Phase 2 (Experimental): Subjects aged ≥60 years in phase 2 will receive single dose of Recombinant Respiratory Syncytial Virus Vaccine (CHO Cells)(low dose), by IM injection into the deltoid region of the arm.
  Interventions: Biological: Recombinant Respiratory Syncytial Virus Vaccine (CHO Cells)(low dose)
- High dose vaccine group in subjects aged ≥60 years - Phase 2 (Experimental): Subjects aged ≥60 years in phase 2 will receive single dose of Recombinant Respiratory Syncytial Virus Vaccine (CHO Cells)(high dose), by IM injection into the deltoid region of the arm.
  Interventions: Biological: Recombinant Respiratory Syncytial Virus Vaccine (CHO Cells)(high dose)
- Placebo group in subjects aged ≥60 years - Phase 2 (Placebo Comparator): Subjects aged ≥60 years in phase 2 will receive single dose of placebo, by IM injection into the deltoid region of the arm.
  Interventions: Biological: Placebo (Saline solution)

INTERVENTIONS:
Biological: Recombinant Respiratory Syncytial Virus Vaccine (CHO Cells)(low dose) — 0.25 mL per dose.
  Arms: Low dose vaccine group in subjects aged 18-59 years - Phase 1; Low dose vaccine group in subjects aged 50-59 years - Phase 2; Low dose vaccine group in subjects aged ≥60 years - Phase 1; Low dose vaccine group in subjects aged ≥60 years - Phase 2
Biological: Recombinant Respiratory Syncytial Virus Vaccine (CHO Cells)(high dose) — 0.5 mL per dose
  Arms: High dose vaccine group in subjects aged 18-59 years - Phase 1; High dose vaccine group in subjects aged 50-59 years - Phase 2; High dose vaccine group in subjects aged ≥60 years - Phase 1; High dose vaccine group in subjects aged ≥60 years - Phase 2
Biological: Placebo (Saline solution) — 0.5 mL per dose
  Arms: Placebo group in subjects aged 18-59 years - Phase 1; Placebo group in subjects aged 50-59 years - Phase 2; Placebo group in subjects aged ≥60 years - Phase 1; Placebo group in subjects aged ≥60 years - Phase 2

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity of two dose levels of the single dose Recombinant RSV vaccine(CHO cells), when administered intramuscularly (IM) in healthy adults aged 18 years and older.

DETAILED DESCRIPTION:
A total of 522 subjects in the phase 1/2 study will be enrolled. The study will be conducted in 2 parts (phase 1 for dose escalation and phase 2 for expansion), with first evaluation of safety of 2 two dose levels of Recombinant RSV vaccine(CHO cells) in healthy participants aged 18-59 and ≥60 in phase 1 before preceding with vaccination of the participants aged 50-59 and ≥60 in phase 2. To ensure the safety of the study participants, phase 1 will follow a staggered enrolment with 3 steps. All subjects in each age group in phase 1 will be randomly receive the investigational vaccine(half or full dose) and the placebo in a 2:1 ratio, while all subjects in each age group in phase 2 will be randomly receive the half dose vaccine, the full dose vaccine and the placebo in a 1:1:1 ratio.

ELIGIBILITY:
Inclusion Criteria:

1. A male or female, in the opinion of the investigator, aged 18 and older for phase 1 and aged 50 and older for phase 2 at the time of the enrollment;
2. Be able to understand the trial procedures, risks and benefits and voluntarily agree to participate in the study and signed an informed consent;
3. Be able to participate in all scheduled visits and comply with the protocol requirements;
4. Women of childbearing potential are willing to use effective contraception (e.g. oral contraceptives, injectable progestogen, implants of levonorgestrel, percutaneous contraceptive patches, intrauterine device (IUD), female and male sterilization, abstinence, condoms, or diaphragms), and the rhythm method, withdrawal and emergency contraception pills are not acceptable;
5. Subjects with stable conditions considered by the investigator.

Exclusion Criteria:

1. Axillary temperature>37.0℃;
2. History of RSV infection within 6 months before enrollment;
3. New onset of respiratory tract infection symptoms like cough, sputum, shortness of breath, wheezing, fever, runny nose or nasal congestion within 7 days before enrollment;
4. Acute diseases or acute exacerbation of chronic disease within 3 days before vaccination;
5. A known allergy to any components of the study vaccine, or history of severe allergy (e.g. anaphylactic shock, allergic laryngeal edema, anaphylactoid purpura, thrombocytopenic purpura, Arthus reaction, severe urticaria) or serious adverse reactions to any previous vaccination or drug use;
6. Pregnant (urine pregnancy test was positive) or lactating female, or planned pregnancy within 12 months after vaccination;
7. Any confirmed or suspected immunosuppressive or immunodeficient condition due to diseases or immunosuppressive therapy, based on medical history and physical examination;
8. Serious or unstable chronic illness, including but not limit to cardiovascular diseases (such as uncontrolled hypertension, coronary heart disease, myocarditis, pericarditis), metabolic diseases (such as poorly controlled diabetes), hematological diseases (such as severe anemia, hemophilia), liver and kidney diseases, digestive diseases, respiratory diseases (such as chronic obstructive pulmonary disease, active tuberculosis, other severe respiratory diseases ), malignant tumor, major functional organ transplantation history;
9. Significant underlying illness that in the opinion of the investigator would be expected to prevent completion of the study;
10. History of thrombocytopenia or other coagulation disorders;
11. History of convulsions, epilepsy, congenital brain dysplasia, mental illness or family history, or history of brain nerve tissue damage due to other severe neurological disorders(e.g. brain tumor, cerebral hemorrhage, cerebral infarction, brain infection disease, chemical drug poisoning);
12. History of cognitive dysfunction, or any moderate or severe cognitive impairment;
13. Asplenia or functional asplenia, or autoimmune thyroid diseases, such as Hashimoto thyroiditis, toxic diffuse goiter;
14. Receipt of live vaccine within 28 days, or any other vaccine within 14 days prior to vaccination;
15. Previous vaccination with an RSV vaccine;
16. Administration of long-acting immune-modifying drugs(e.g. Infliximab) or planned administration at any time during the study period;
17. Administration of immunoglobulins and/or any blood products during the period starting 3 months before vaccination or planned administration during the study period;
18. Chronic administration of immunosuppressants or other immune-modifying drugs (such as long-term use of systemic glucocorticoid ≥14 days, ≥20mg/day prednisone or equivalent dose) during the period starting 3 months before vaccination or planned administration during the study period, but topical steroids(e.g. ointment, eye drops, inhalants, nasal sprays) that do not exceed the dosage recommended in the instructions or have any systemic signs are acceptable;
19. History of alcohol or drug abuse;
20. Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational vaccine/product;
21. Planned move to a location that will prohibit participating in the trial until study end;
22. At screening: Any laboratory test results(hematology, clinical chemistry, coagulation function, or urinalysis) abnormal and clinically significant in the judgment of the investigator (Only for phase 1);
23. At screening: Any electrocardiogram abnormal and clinically significant in the judgment of the investigator (Only for phase 1);
24. Any condition that, in the opinion the investigator, may affect the safety of the subject or the evaluation of the study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 522 (Estimated)
Dates: Start 2024-11-13 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
Incidence, Intensity and Causality of adverse events(AE) | Within 30 days after vaccination
  An AE includes any untoward medical occurrence in a patient or clinical investigation subject administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. An AE can therefore be any unfavourable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a investigational product, whether or not related to the investigational product.
Incidence, Intensity and Causality of solicited AEs | Within 14 days after vaccination
  Solicited AEs include solicited local and general symptoms; Assessed solicited local AEs at injection site are pain, erythema, swelling, induration and itching; Assessed solicited general symptoms include fever, fatigue, headache, myalgia, nausea, vomiting, diarrhea, arthralgia and hypersensitivity.
Incidence, Intensity and Causality of unsolicited AEs | Within 30 days after vaccination
  An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and/or any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Incidence, Intensity and Causality of Severe adverse events(SAEs) | Within 30 days after vaccination
  SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in persistent or significant disability/incapacity or are congenital anomaly/birth defect.
Incidence, Intensity and Causality of Adverse events of special interest(AESI) | Within 30 days after vaccination
  Adverse events of special interest include potential immune-mediated diseases and atrial fibrillation.
Incidence of abnormal and clinically significant laboratory test results - only for phase 1 | The 3rd day after vaccination
  Laboratory test includes hematology, blood biochemistry, coagulation test, urine analysis and Electrocardiograph.
Geometric Mean Titer (GMT) of Neutralizing Antibody against RSV-serotype A | 30 days after vaccination
  Measured by Virus Neutralization Test.
GMT of Neutralizing Antibody against RSV-serotype B | 30 days after vaccination
  Measured by Virus Neutralization Test.
Geometric Mean Fold Rise (GMFR) of Neutralizing Antibody against RSV-serotype A | 30 days after vaccination
  Compared with the baseline Titer(Day 0).
GMFR of Neutralizing Antibody against RSV-serotype B | 30 days after vaccination
  Compared with the baseline Titer(Day 0).
Geometric Mean Concentration (GMC) of RSV-Prefusion F protein(RSV-PreF) specific Immunoglobulin G (IgG) Antibody against RSV-serotype A | 30 days after vaccination
  Measured by ELISA.
GMC of RSV-PreF specific IgG Antibody against RSV-serotype B | 30 days after vaccination
  Measured by ELISA.
GMFR of RSV-PreF specific IgG Antibody against RSV-serotype A | 30 days after vaccination
  Compared with the baseline concentration(Day 0).
GMFR of RSV-PreF specific IgG Antibody against RSV-serotype B | 30 days after vaccination
  Compared with the baseline concentration(Day 0).

SECONDARY OUTCOMES:
Incidence, Intensity and Causality of SAEs | Up to 12 months post vaccination
  SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in persistent or significant disability/incapacity or are congenital anomaly/birth defect.
Incidence, Intensity and Causality of AESI | Up to 12 months post vaccination
  Adverse events of special interest include potential immune-mediated diseases and atrial fibrillation.
GMT of Neutralizing Antibody against RSV-serotype A and RSV-serotype B | 14 days post vaccination-only for phase 1
  Measured by Virus Neutralization Test.
GMFR of Neutralizing Antibody against RSV-serotype A and RSV-serotype B | 14 days post vaccination-only for phase 1
  Compared with the baseline Titer(Day 0).
GMC of RSV-PreF specific IgG Antibody against RSV-serotype A and RSV-serotype B | 14 days post vaccination-only for phase 1
  Measured by ELISA.
GMFR of RSV-PreF specific IgG Antibody against RSV-serotype A and RSV-serotype B | 14 days post vaccination-only for phase 1
  Compared with the baseline concentration(Day 0).
GMT of Neutralizing Antibody against RSV-serotype A and RSV-serotype B | At 6, 12, and 24 months post vaccination
  Measured by Virus Neutralization Test.
GMFR of Neutralizing Antibody against RSV-serotype A and RSV-serotype B | At 6, 12, and 24 months post vaccination
  Compared with the baseline Titer(Day 0).
GMC of RSV-PreF specific IgG Antibody against RSV-serotype A and RSV-serotype B | At 6, 12, and 24 months post vaccination
  Measured by ELISA.
GMFR of RSV-PreF specific IgG Antibody against RSV-serotype A and RSV-serotype B | At 6, 12, and 24 months post vaccination
  Compared with the baseline concentration(Day 0).
The Frequency of RSV-PreF Specific Cluster of Differentiation 4+ (CD4+) T Cells or Cluster of Differentiation 8+ (CD8+) T cells Expressing at Least 2 Markers - only for phase 2 | 30 days post vaccination
  Among markers expressed were interleukin-2 (IL-2), cluster of 40 ligand (CD40L), tumor necrosis factor alpha (TNF α) and interferon gamma (IFN γ), in vitro upon stimulation with RSV-PreF peptide preparations.

CONTACTS AND LOCATIONS:
Overall Officials: Lili Huang, Principal Investigator — Henan Center for Disease Control and Prevention
Locations (1):
- Liangyuan District Center for Disease Prevention and Control, Shangqiu, Henan, China

IPD SHARING:
Plan to Share IPD: No